CLINICAL TRIAL: NCT01273155
Title: Phase I Pharmacokinetic Study of Belinostat for Solid Tumors and Lymphomas in Patients With Varying Degrees of Hepatic Dysfunction
Brief Title: Belinostat for Solid Tumors and Lymphomas in Patients With Varying Degrees of Hepatic Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Naoko Takebe, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110060; 11-C-0060
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Neoplasms; Lymphomas
Keywords: Histone Deacetylase Inhibitor; Liver Dysfunction; Pharmacokinetics; UGT1A1 Polymorphisms; Solid Tumor; Cancer; Lymphoma
MeSH Terms: conditions — Neoplasms; Lymphoma; Liver Diseases | interventions — belinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Normal Function-Belinostat 1000 mg/m(2) (Active Comparator): Normal Liver Function was defined as bilirubin ≤Upper Limit of Normal (ULN) and aspartate aminotransferase (AST) ≤ ULN.
  Interventions: Drug: Belinostat
- Mild Dysfunction-Belinostat 750 mg/m(2) (Experimental): Mild Liver Dysfunction was defined as bilirubin >Upper Limit of Normal (ULN) but ≤1.5 x ULN and/or aspartate aminotransferase (AST) > ULN.
  Interventions: Drug: Belinostat
- Mild Dysfunction-Belinostat 1000 mg/m(2) (Experimental): Mild Liver Dysfunction was defined as bilirubin >Upper Limit of Normal (ULN) but ≤1.5 x ULN and/or aspartate aminotransferase (AST) > ULN.
  Interventions: Drug: Belinostat
- Moderate Dysfunction-Belinostat 500 mg/m(2) (Experimental): Moderate Liver Dysfunction was defined as bilirubin >1.5 to ≤ 3 x ULN and any aspartate aminotransferase (AST).
  Interventions: Drug: Belinostat
- Moderate Dysfunction-Belinostat 750 mg/m(2) (Experimental): Moderate Liver Dysfunction was defined as bilirubin >1.5 to ≤ 3 x ULN and any aspartate aminotransferase (AST).
  Interventions: Drug: Belinostat
- Severe Dysfunction-Belinostat 250 mg/m(2) (Experimental): Severe Liver Dysfunction was defined as bilirubin >3 but ≤ 10 x ULN and any aspartate aminotransferase (AST).
  Interventions: Drug: Belinostat
- Severe Dysfunction-Belinostat 350 mg/m(2) (Experimental): Severe Liver Dysfunction was defined as bilirubin >3 but ≤ 10 x ULN and any aspartate aminotransferase (AST).
  Interventions: Drug: Belinostat

INTERVENTIONS:
Drug: Belinostat — Belinostat was administered intravenously (IV) over 30 minutes on days 1 through 5 of a 21-day cycle. All patients were administered a single dose of 400 mg/m(2) of belinostat on Cycle 1 Day -7 for pharmacokinetic analysis (the total length of Cycle 1 was 28 days).
  Other Names: Beleodaq

SUMMARY:
Background:

- Belinostat is an experimental cancer treatment drug that works by helping to turn on genes that limit cell growth and survival of cancer cells. These genes are often switched off in tumors. Belinostat has been given to patients with different types of cancer to measure its safety and effectiveness, but it has not been given in a formal trial to cancer patients who have abnormal liver function. Because belinostat is processed by the liver, its safety and effectiveness needs to be established in individuals who have abnormal liver function. Researchers are interested in comparing the effects of belinostat as a cancer treatment drug in individuals with normal and abnormal liver function.

Objectives:

* To test the safety and effectiveness of belinostat in individuals who have solid tumors and lymphomas and who also have abnormal liver function.
* To compare the results of belinostat treatment in individuals with normal and abnormal liver function.

Eligibility:

* Individuals at least 18 years of age who have been diagnosed with solid tumors or lymphomas that have not responded to standard treatment.
* Individuals with normal liver function and varying degrees of abnormal liver function (mild, moderate, severe) are eligible.

Design:

* Participants will be screened with a full medical history and physical examination, as well as blood and urine tests, and tumor imaging studies. Participants will then be divided into study groups based on their liver function.
* Participants will receive belinostat in cycles of treatment. Except for cycle 1, all cycles will last 21 days. Cycle 1 will last 28 days. For cycle 1 only, participants will receive a single dose of belinostat 1 week before the regular 21-day treatment cycle starts.
* In each cycle, participants will receive belinostat once a day for 5 days, and will be asked to keep a medication diary to record any side effects.
* Participants will have regular clinic visits with blood and urine sample collection and imaging studies to evaluate the cancer's response to treatment.
* Participants may continue to take belinostat for as long as the cancer responds to the treatment.

DETAILED DESCRIPTION:
Background:

* Belinostat is a histone deacetylase (HDAC) inhibitor. HDACs are frequently deregulated in cancer cells, leading to an increase in deacetylation and the silencing of genes that normally control cell cycle arrest and apoptosis.
* Belinostat has growth inhibitory activity in several malignancies in vitro and in vivo, both as a single agent and in combination with chemotherapeutic agents. Several Phase I and II clinical trials have been conducted to date in patients with solid tumor and hematologic malignancies; belinostat has been generally well tolerated.
* Belinostat is metabolized in the liver and therefore, the safety and dosing of belinostat needs to be established in patients with varying degrees of hepatic dysfunction.

Objectives:

* Establish the safety and tolerability of belinostat given on days 1 through 5 of 21-day cycles to patients with varying degrees of liver dysfunction.
* Define the maximum tolerated dose (MTD) and recommended dose of belinostat given on days 1 through 5 of 21-day cycles to patients with varying degrees of liver dysfunction.
* Evaluate the pharmacokinetics (PK) of one dose of belinostat (400 mg/m(2)) in patients with varying degrees of liver dysfunction.
* Obtain preliminary evidence of anti-tumor activity at tolerable doses of belinostat in patients with varying degrees of liver dysfunction.
* Measure direct versus indirect bilirubin levels and correlate these with observed toxicities, PK.

Eligibility:

-Adults with solid tumors or lymphomas whose disease has progressed after standard therapy or who have no acceptable standard treatment options. Patients with normal and varying degrees of hepatic dysfunction (mild, moderate, and severe) are eligible.

Study Design:

-Patients will be divided into 4 dose escalation cohorts based on their level of liver dysfunction. Belinostat will be administered intravenously (IV) over 30 minutes. On day -7 (Cycle 1 only), all patients will receive a single dose of 400 mg/m(2) belinostat. On days 1 through 5 of each cycle, patients will receive belinostat at a dose dependent on the level of hepatic dysfunction and dose level. Mild, moderate, and severe liver dysfunction cohorts will begin on dose level 1; patients with normal hepatic function will not have their dose escalated (see below). The total length of Cycle 1 will be 28 days; all other cycles will be 21 days. No more than 12 evaluable patients with normal hepatic function will be accrued.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients must have histologically or cytologically confirmed (at original diagnosis or subsequent recurrence or progression) solid tumor or lymphoma that is metastatic, unresectable, progressive, or recurrent, and for which standard curative or palliative measures do not exist or are no longer effective.
* No radiation, major surgery, chemotherapy or biologic therapy within 4 weeks prior to entering the study (6 weeks for nitrosoureas or mitomycin C); greater than or equal to 2 weeks since any prior administration of study drug in an exploratory Investigational New Drug (IND)/Phase 0 study. (also referred to as an "early Phase I study" or "pre-Phase I study" where a sub-therapeutic dose of drug is administered) at the Principal Investigator's (PI's) discretion. Patients must have recovered to at least eligibility levels due to adverse events and/or toxicity of prior chemotherapy or biologic therapy.
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of belinostat in patients < 18 years of age, children are excluded from this study but will be eligible for future pediatric Phase I single-agent trials.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 (Karnofsky greater than or equal to 60 percent.
* Life expectancy of greater than 3 months.
* Patients must have acceptable renal and marrow function as defined below:

leukocytes greater than or equal to 3,000/mcL

absolute neutrophil count greater than or equal to 1,500/mcL

platelets greater than or equal to 100,000/mcL

serum creatinine within normal institutional limits OR creatinine clearance greater than or equal to 60 mL/min for patients with creatinine levels above institutional normal, as determined by a measured 24-hour creatinine clearance Baseline evaluations should be conducted within 7 days of treatment start date.

* Patients with abnormal liver function will be eligible. Patients with active hemolysis should be excluded. No distinction will be made between liver dysfunction due to metastases and liver dysfunction due to other causes.
* Patients with biliary obstruction for which a stent has been placed are eligible, provided the stent has been in place for at least 10 days prior to the first dose of belinostat and the liver function has stabilized. Two measurements at least 2 days apart that put the patient in the same hepatic dysfunction stratum will be accepted as evidence of stable hepatic function. There should be no evidence of biliary sepsis.
* Patients with gliomas or brain metastases who require corticosteroids or anticonvulsants must be on a stable dose of corticosteroids and seizure free for 1 month prior to enrollment. Patients with known brain metastases should have had brain irradiation (whole brain or gamma knife) more than 4 weeks before starting the protocol. Note that patients should have had their steroids tapered to low dose (i.e., < 1.5 mg of dexamethasone/day).
* The effects of belinostat on the developing human fetus are unknown. For this reason and because histone deacetylase (HDAC) inhibitors are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Prior therapy with belinostat.
* Patients may not be receiving any other investigational agents.
* Patients with history of allergic reactions attributed to compounds of similar chemical or biologic composition to belinostat, including hydroxamate compounds or arginine.
* Patients should not have taken valproic acid, another HDAC inhibitor, for at least 2 weeks prior to enrollment.
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because belinostat is an HDAC inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with belinostat, breastfeeding should be discontinued if the mother is treated with belinostat.
* Human Immunodeficiency Virus (HIV) positive patients who are not on retroviral therapy will not be excluded from cohort 1, the normal liver function cohort. HIV positive patients who are not on retroviral therapy will be excluded from cohorts 2-4 because of confounding effects from potential complications from HIV and opportunistic infections.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for the increased risk of liver dysfunction from the antiretroviral therapies themselves and because of potential pharmacokinetics (PK) interactions with belinostat. Appropriate studies will be undertaken in these groups of patients when indicated.
* Patients with significant cardiovascular disease (New York Heart Association Class III or IV cardiac disease), symptomatic congestive heart failure, myocardial infarction within the past 6 months, unstable angina, unstable arrhythmia or a need for anti-arrhythmic therapy (use of frequency adjusting medication for atrial fibrillation is allowed, if stable medication for at least last month prior to initiation of belinostat treatment and medication not listed as causing Torsades de Points), or evidence of acute ischemia on electrocardiogram (ECG). Marked baseline prolongation of Q wave, T wave (QT)/Corrected QT Interval (QTc) interval, e.g., repeated demonstration of a QTc interval > 450 msec; Long QT Syndrome; the required use of concomitant medication that may cause Torsades de Pointes.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-01-10 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoko Takebe, M.D., Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (7):
- United States (7):
  - University of California, Davis, Davis, California
  - City of Hope National Medical Center, Duarte, California
  - USC Norris Cancer Center, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Albert Einstein College of Medicine, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Plumb JA, Finn PW, Williams RJ, Bandara MJ, Romero MR, Watkins CJ, La Thangue NB, Brown R. Pharmacodynamic response and inhibition of growth of human tumor xenografts by the novel histone deacetylase inhibitor PXD101. Mol Cancer Ther. 2003 Aug;2(8):721-8. PMID 12939461
- [Background] Gimsing P. Belinostat: a new broad acting antineoplastic histone deacetylase inhibitor. Expert Opin Investig Drugs. 2009 Apr;18(4):501-8. doi: 10.1517/13543780902852560. PMID 19335278
- [Background] Marks PA, Richon VM, Rifkind RA. Histone deacetylase inhibitors: inducers of differentiation or apoptosis of transformed cells. J Natl Cancer Inst. 2000 Aug 2;92(15):1210-6. doi: 10.1093/jnci/92.15.1210. PMID 10922406
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0060.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Function-Belinostat 1000 mg/m(2) | Mild Dysfunction-Belinostat 750 mg/m(2) | Mild Dysfunction-Belinostat 1000 mg/m(2) | Moderate Dysfunction-Belinostat 500 mg/m(2) | Moderate Dysfunction-Belinostat 750 mg/m(2) | Severe Dysfunction-Belinostat 250 mg/m(2) | Severe Dysfunction-Belinostat 350 mg/m(2)
Started | 14 | 12 | 18 | 5 | 5 | 10 | 8
Completed | 12 | 8 | 6 | 4 | 3 | 5 | 2
Not Completed | 2 | 4 | 12 | 1 | 2 | 5 | 6
Not completed — Off study trmt prior to end of C1/PD | 2 | 3 | 8 | 0 | 0 | 2 | 3
Not completed — Change in liver function/no longer eval. | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Off study prior to C1/due to toxicity | 0 | 0 | 2 | 0 | 0 | 0 | 1
Not completed — Died during Cycle 1 | 0 | 0 | 1 | 1 | 0 | 2 | 2
Not completed — Withdrew during C1/refused further trmt | 0 | 0 | 1 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Normal Function: Normal Liver Function was defined as bilirubin ≤Upper Limit of Normal (ULN) and aspartate aminotransferase (AST) ≤ ULN.
  Belinostat: Belinostat was administered intravenously (IV) over 30 minutes on days 1 through 5 of a 21-day cycle. All patients were administered a single dose of 400 mg/m(2) of belinostat on Cycle 1 Day -7 for pharmacokinetic analysis (the total length of Cycle 1 was 28 days).
- Mild Dysfunction: Mild Liver Dysfunction was defined as bilirubin >Upper Limit of Normal (ULN) but ≤1.5 x ULN and/or aspartate aminotransferase (AST) > ULN.
  Belinostat: Belinostat was administered intravenously (IV) over 30 minutes on days 1 through 5 of a 21-day cycle. All patients were administered a single dose of 400 mg/m(2) of belinostat on Cycle 1 Day -7 for pharmacokinetic analysis (the total length of Cycle 1 was 28 days).
- Moderate Dysfunction: Moderate Liver Dysfunction was defined as bilirubin >1.5 to ≤ 3 x ULN and any aspartate aminotransferase (AST).
  Belinostat: Belinostat was administered intravenously (IV) over 30 minutes on days 1 through 5 of a 21-day cycle. All patients were administered a single dose of 400 mg/m(2) of belinostat on Cycle 1 Day -7 for pharmacokinetic analysis (the total length of Cycle 1 was 28 days).
- Severe Dysfunction: Severe Liver Dysfunction was defined as bilirubin >3 but ≤ 10 x ULN and any aspartate aminotransferase (AST).
  Belinostat: Belinostat was administered intravenously (IV) over 30 minutes on days 1 through 5 of a 21-day cycle. All patients were administered a single dose of 400 mg/m(2) of belinostat on Cycle 1 Day -7 for pharmacokinetic analysis (the total length of Cycle 1 was 28 days).
- Total: Total of all reporting groups
Arm/Group | Normal Function | Mild Dysfunction | Moderate Dysfunction | Severe Dysfunction | Total
Number analyzed (Participants) | 14 | 30 | 10 | 18 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 22 | 6 | 12 | 47
  >=65 years | 7 | 8 | 4 | 6 | 25
Age, Continuous [Median (Full Range); unit: years] | 65 [46 to 73] | 59 [30 to 73] | 63.5 [53 to 73] | 57.5 [35 to 77] | 61 [30 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 3 | 8 | 28
  Male | 8 | 19 | 7 | 10 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3 | 6
  Not Hispanic or Latino | 13 | 29 | 9 | 15 | 66
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 8 | 2 | 2 | 16
  White | 10 | 19 | 8 | 15 | 52
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 30 | 10 | 18 | 72
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — Gr 0: Fully active, able to carry on all pre-disease performance without restriction.
  Gr 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Gr 2: Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Gr 3: Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours.
  Gr 4: Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Gr 5: Dead.
  Participants
    Grade 0 | 4 | 2 | 3 | 1 | 10
    Grade 1 | 9 | 26 | 5 | 13 | 53
    Grade 2 | 1 | 2 | 2 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLTs)
Description: A DLT was defined as an adverse event deemed possibly, probably, or definitely related to administration of study drugs and met the following criteria: grade≥3 non-hematological toxicity (except grade ≥3 diarrhea, nausea, vomiting responsive to supportive therapy);grade≥3 rise in creatinine (except grade 3 able to be corrected to grade 1 or baseline with intravenous fluids within 24hrs); grade≥3 electrolyte toxicities (except those able to be corrected to grade 1 or baseline within 48hrs); grade 4 thrombocytopenia; grade 4 neutropenia for >5 days or febrile neutropenia; any neurotoxicity grade≥2 not reversible to grade 1 or baseline within 2wks; or any delay in treatment by ≥2wks due to treatment-related toxicity. Worsening liver function, as defined by a rise in serum bilirubin not related to tumor progression, was considered a DLT if a patient with mild dysfunction became severe for 1wk, or if a patient in either the moderate/severe groups had a >1.5x increase in bilirubin for 1 wk.
Time Frame: First cycle of therapy, 28 days.
Population: Forty patients were evaluable for dose-limiting toxicity; others came off study prior to the end of Cycle 1 and were not evaluable.
Measure: Number; unit: Toxicities
Arm/Group | Normal Function-Belinostat 1000 mg/m(2) | Mild Dysfunction-Belinostat 750 mg/m(2) | Mild Dysfunction-Belinostat 1000 mg/m(2) | Moderate Dysfunction-Belinostat 500 mg/m(2) | Moderate Dysfunction-Belinostat 750 mg/m(2) | Severe Dysfunction-Belinostat 250 mg/m(2) | Severe Dysfunction-Belinostat 350 mg/m(2)
Number analyzed (Participants) | 12 | 8 | 6 | 4 | 3 | 5 | 2
Toxicities | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Belinostat According to Degree of Liver Dysfunction
Description: In order to maintain consistent dosing across the hepatic dysfunction groups, the dose recommended for cohorts with greater liver dysfunction could be no greater than the dose for cohorts of lesser dysfunction. In other words, it was assumed that a particular group would not tolerate a dose not tolerated by a group with lesser dysfunction and conversely, will tolerate a dose tolerated by a group with greater dysfunction. If a higher dose was tolerated in a group of greater dysfunction, but not in the group of lesser dysfunction, the lower dose would be recommended for both groups. The highest dose to be explored was no greater than the recommended dose for patients with normal liver function.
Time Frame: First cycle of therapy, 28 days
Population: Normal liver function patients were not eligible for dose escalation. Twenty-eight patients were evaluable for MTD; others came off study prior to the end of Cycle 1 and were not evaluable.
Measure: Number; unit: mg/m(2)
Arm/Group | Mild Dysfunction | Moderate Dysfunction | Severe Dysfunction
Number analyzed (Participants) | 14 | 7 | 7
mg/m(2) | 1000 | NA — The MTD was not established for the moderate and severe cohorts prior to study closure. | NA — The MTD was not established for the moderate and severe cohorts prior to study closure.

3. Primary Outcome: Number of Participants Experiencing Adverse Events Considered to be at Least Possibly Related to the Study Drug
Description: The number of participants experiencing each adverse event by liver function cohort at each dose level. The grade refers to the severity of the Adverse Event. Grade 1 Mild; Grade 2 Moderate; Grade 3 Severe or medically significant but not immediately life-threatening; Grade 4 Life-threatening consequences; Grade 5 Death related to adverse event.
Time Frame: From Cycle 1 Day -7 up to 12 (21-day) cycles
Population: Total number of evaluable patients per cohort on the indicated dose level; only patients who received study drug were evaluable for assessment of toxicity (some patients were assigned to a dose level but did not receive study drug and are therefore not included).
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Function-Belinostat 1000 mg/m(2) | Mild Dysfunction-Belinostat 750 mg/m(2) | Mild Dysfunction-Belinostat 1000 mg/m(2) | Moderate Dysfunction-Belinostat 500 mg/m(2) | Moderate Dysfunction-Belinostat 750 mg/m(2) | Severe Dysfunction-Belinostat 250 mg/m(2) | Severe Dysfunction-Belinostat 350 mg/m(2)
Number analyzed (Participants) | 14 | 10 | 15 | 5 | 6 | 9 | 5
Participants
  Grade 2 Anemia | 1 | 1 | 3 | 0 | 1 | 0 | 1
  Grade 3 Anemia | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 Anorexia | 1 | 0 | 1 | 1 | 0 | 0 | 0
  Grade 2 Dyspepsia | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Dyspnea | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Edema (limbs) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Fatigue | 2 | 1 | 2 | 1 | 1 | 1 | 0
  Grade 3 Fatigue | 1 | 1 | 2 | 0 | 2 | 0 | 0
  Grade 2 Hypertension | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 Hypophosphatemia | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 Hypophosphatemia | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Infusion related reaction | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 2 infusion site extravasation | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 INR Increased | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5 Lung Infection | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 Lymphocyte count decreased | 1 | 0 | 4 | 1 | 1 | 0 | 1
  Grade 3 Lymphocyte count decreased | 3 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Nausea | 3 | 0 | 3 | 0 | 0 | 0 | 0
  Grade 3 Pain in extremity | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 Peripheral nerve infection | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 Phlebitis | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 Rash maculo-papular | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 3 Syncope | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 Vomiting | 1 | 1 | 1 | 0 | 0 | 1 | 0
  Grade 3 Vomiting | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Weight loss | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 White blood cell decreased | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 Abdominal distension | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Alanine aminotransferase increased | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Grade 3 Ascites | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Aspartate aminotransferase increased | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Grade 2 Blood bilirubin increased | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Blood bilirubin increased | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Grade 4 Blood bilirubin increased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Chills | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Constipation | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Diarrhea | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Fever | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 Generalized muscle weakness | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Infections and infestations - Other | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Malaise | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Platelet count decreased | 0 | 0 | 0 | 0 | 1 | 0 | 0

4. Primary Outcome: Pharmacokinetics (PK) of a Single-dose Belinostat (400 mg/m^2)) According to Degree of Liver Dysfunction: Maximum Plasma Concentrations (Cmax)
Description: Maximum plasma concentrations (Cmax) for belinostat and five metabolites on Cycle 1 Day -7 as a function of degree of liver dysfunction.
Time Frame: Cycle 1 Day -7 prior to infusion; 15 and 25 minutes after the start of infusion; and 5, 10, 15, 30, 60, and 90 minutes, and 2, 4, 6, 8, and 24 hours after the end of infusion.
Population: The number of patients in a given cohort that received Belinistat on Cycle 1 Day-7 and had blood samples successfully collected at the specified timepoints for PK analysis. There were 3 patients with Mild Liver Dysfunction who were not evaluable for Belinostat Cmax.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Normal Function | Mild Dysfunction | Moderate Dysfunction | Severe Dysfunction
Number analyzed (Participants) | 14 | 25 | 10 | 15
µg/mL
  Belinostat: number analyzed (Participants) | 14 | 22 | 10 | 15
  Belinostat | 21.9 (8.7) | 26.6 (9.5) | 22.1 (5.7) | 25.0 (7.4)
  Belinostat glucuronide | 80.8 (27.3) | 90.8 (19.2) | 67.2 (33.6) | 72.8 (28.2)
  Methyl belinostat | 2.10 (0.94) | 2.99 (1.15) | 3.26 (0.75) | 3.35 (0.90)
  M21 | 1.26 (0.75) | 1.79 (0.70) | 1.64 (0.32) | 1.93 (0.59)
  M24 | 2.56 (0.77) | 2.35 (0.96) | 1.82 (0.65) | 1.88 (0.96)
  M26 | 1.68 (0.71) | 1.80 (0.64) | 1.83 (0.52) | 2.24 (1.65)
Statistical Analysis 1: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; Effects of liver dysfunction on PK parameter values were evaluated with SPSS 22.0 for Windows (SPSS Inc., Chicago, IL), using the Jonckheere-Terpstra and Kendall's Tau test. Data were considered significantly different when p<0.05; Test type: Other — Belinostat; p = 0.327, Jonckheere-Terpstra; Kendall's Tau = 0.096
Statistical Analysis 2: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — Belinostat glucuronide; p = 0.063, Jonckheere-Terpstra; Kendall's Tau = -0.178
Statistical Analysis 3: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — Methyl belinostat; p < 0.001, Jonckheere-Terpstra; Kendall's Tau = 0.382
Statistical Analysis 4: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — M21; p = 0.009, Jonckheere-Terpstra; Kendall's Tau = 0.253
Statistical Analysis 5: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — M24; p = 0.004, Jonckheere-Terpstra; Kendall's Tau = -0.278
Statistical Analysis 6: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — M26; p = 0.312, Jonckheere-Terpstra; Kendall's Tau = 0.098

5. Primary Outcome: Pharmacokinetics (PK) of Single-dose Belinostat (400 mg/m^2) According to Degree of Liver Dysfunction: Area Under the Plasma Concentration Time Curve Extrapolated to Infinity(AUC0-inf)
Description: Area Under the Plasma Concentration Time Curve Extrapolated to Infinity (AUC0-inf) for belinostat and four metabolites on Cycle 1 Day -7 as a function of degree of liver dysfunction.
Time Frame: Cycle 1 Day-7 prior to infusion; 15 and 25 minutes after start of infusion; and 5, 10, 15, 60, 60, and 90 minutes, and 2, 4, 6, 8, and 24 hours after the end of infusion.
Population: The number of patients in a given cohort that received Belinostat on Cycle 1 day -7 and had blood samples successfully collected at the specified timepoints for PK analysis. One patient with Mild Liver Dysfunction was not evaluated for Belinostat AUC0-inf.
Measure: Mean (Standard Deviation); unit: µg*min/mL
Arm/Group | Normal Function | Mild Dysfunction | Moderate Dysfunction | Severe Dysfunction
Number analyzed (Participants) | 14 | 25 | 10 | 15
µg*min/mL
  Belinostat: number analyzed (Participants) | 14 | 24 | 10 | 15
  Belinostat | 719 (265) | 859 (270) | 834 (217) | 1012 (408)
  Methyl belinostat | 354 (305) | 483 (163) | 829 (471) | 930 (797)
  M21 | 647 (884) | 840 (589) | 1058 (398) | 1295 (600)
  M24 | 1009 (555) | 916 (450) | 885 (514) | 970 (693)
  M26 | 361 (193) | 396 (164) | 600 (292) | 740 (576)
Statistical Analysis 1: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — Belinostat; p = 0.025, Jonckheere-Terpstra; Kendall's Tau = 0.215
Statistical Analysis 2: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — Methyl belinostat; p < 0.001, Jonckheere-Terpstra; Kendall's Tau = 0.426
Statistical Analysis 3: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — M21; p < 0.001, Jonckheere-Terpstra; Kendall's Tau = 0.337
Statistical Analysis 4: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — M24; p = 0.524, Jonckheere-Terpstra; Kendall's Tau = -0.061
Statistical Analysis 5: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — M26; p = 0.010, Jonckheere-Terpstra; Kendall's Tau = 0.246

6. Primary Outcome: Pharmacokinetics (PK) of Single-dose Belinostat (400 mg/m^2) According to Degree of Liver Dysfunction: Area Under the Plasma Concentration Time Curve Extrapolated to Infinity(AUC0-inf) of Belinostat
Description: Area Under the Plasma Concentration Time Curve Extrapolated to Infinity(AUC0-inf) for Belinostat glucuronide, a Belinostat Metabolite on Cycle 1 Day-7 as a function of degree of liver dysfunction.
Time Frame: as for outcome 4
Population: The number of patients in a given cohort that received Belinostat on Cycle 1 Day -7 and had blood samples successfully collected at the specified timepoints for PK analysis.
Measure: Mean (Standard Deviation); unit: mg*min/mL
Arm/Group | Normal Function | Mild Dysfunction | Moderate Dysfunction | Severe Dysfunction
Number analyzed (Participants) | 14 | 25 | 10 | 15
mg*min/mL | 15.1 (10.4) | 18.4 (5.9) | 18.4 (13.4) | 23.4 (25.6)
Statistical Analysis 1: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.548, Jonckheere-Terpstra; Kendall's Tau = 0.057

7. Primary Outcome: Pharmacokinetics (PK) of Single-dose Belinostat (400 mg/m^2) According to Degree of Liver Dysfunction: Half-Life (t1/2)
Description: Half-life Period (t1/2) of belinostat and five metabolites on Cycle 1 Day -7 as a function of degree of liver function.
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Normal Function | Mild Dysfunction | Moderate Dysfunction | Severe Dysfunction
Number analyzed (Participants) | 14 | 25 | 10 | 15
min
  Belinostat | 118 (90) | 127 (57) | 144 (86) | 157 (118)
  Belinostat glucuronide | 280 (55) | 246 (59) | 238 (128) | 267 (134)
  Methyl belinostat | 79.6 (38.9) | 80.3 (19.1) | 136.1 (96.0) | 133 (98)
  M21 | 305 (337) | 460 (324) | 486 (191) | 485 (205)
  M24 | 264 (106) | 253 (97) | 223 (119) | 260 (133)
  M26 | 131 (115) | 151 (194) | 177 (95) | 153 (83)
Statistical Analysis 1: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — Belinostat; p = 0.340, Jonckheere-Terpstra; Kendall's Tau = 0.091
Statistical Analysis 2: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — Belinostat glucuronide; p = 0.023, Jonckheere-Terpstra; Kendall's Tau = -0.216
Statistical Analysis 3: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — Methyl belinostat; p = 0.005, Jonckheere-Terpstra; Kendall's Tau = 0.268
Statistical Analysis 4: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — M21; p = 0.011, Jonckheere-Terpstra; Kendall's Tau = 0.242
Statistical Analysis 5: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — M24; p = 0.231, Jonckheere-Terpstra; Kendall's Tau = -0.114
Statistical Analysis 6: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — M26; p = 0.021, Jonckheere-Terpstra; Kendall's Tau = 0.220

8. Primary Outcome: Pharmacokinetics (PK) of Single-dose Belinostat (400 mg/m^2) According to Degree of Liver Dysfunction: Clearance (CL)
Description: Clearance (CL) of Belinostat on Cycle 1 Day-7 as a function of degree of liver dysfunction
Time Frame: Cycle 1 Day-7 prior to infusion; 15 and 25 minutes after the start of infusion; and 5, 10, 15, 30, 60, and 90 minutes, and 2, 4, 6, 8, and 24 hours after the end of infusion.
Population: The number of patients in a given cohort that received Belinistat on Cycle 1 Day-7 and had blood samples successfully collected at the specified timepoints for PK analysis.
Measure: Mean (Standard Deviation); unit: mL/min/m^2
Arm/Group | Normal Function | Mild Dysfunction | Moderate Dysfunction | Severe Dysfunction
Number analyzed (Participants) | 14 | 25 | 10 | 15
mL/min/m^2 | 661 (346) | 542 (214) | 505 (114) | 444 (137)
Statistical Analysis 1: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.023, Jonckheere-Terpstra; Kendall's Tau = -0.216

9. Primary Outcome: Pharmacokinetics (PK) of Single-dose Belinostat (400 mg/m^2) According to Degree of Liver Dysfunction: Volume of Distribution at Steady State (Vss)
Description: Belinostat Apparent volume of distribution at steady state (Vss) on Cycle 1 Day-7 as a function of degree of liver dysfunction.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: L/m^2
Arm/Group | Normal Function | Mild Dysfunction | Moderate Dysfunction | Severe Dysfunction
Number analyzed (Participants) | 14 | 25 | 10 | 15
L/m^2 | 30.1 (16.1) | 25.7 (17.4) | 38.1 (40.4) | 29.6 (15.4)
Statistical Analysis 1: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.531, Jonckheere-Terpstra; Kendall's Tau = 0.060

10. Primary Outcome: Pharmacokinetics (PK) of Single-dose Belinostat (400 mg/m^2) According to Degree of Liver Dysfunction: Metabolic Ratios of Maximum Plasma Concentrations (Cmax) for the Belinostat Metabolic Pathway
Description: Metabolic ratios of Maximum Plasma Concentrations (Cmax), reported as a geometric mean (geometric standard deviation), for the belinostat metabolic pathway on Cycle 1 Day-7 as a function of degree of liver dysfunction.
Time Frame: as for outcome 8
Population: as for outcome 4
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Normal Function | Mild Dysfunction | Moderate Dysfunction | Severe Dysfunction
Number analyzed (Participants) | 14 | 25 | 10 | 15
ratio
  Belinostat glucuronide/belinostat: number analyzed (Participants) | 14 | 22 | 10 | 15
  Belinostat glucuronide/belinostat | 3.78 (1.47) | 3.57 (1.47) | 2.88 (1.54) | 2.85 (1.51)
  Methyl belinostat/belinostat: number analyzed (Participants) | 14 | 22 | 10 | 15
  Methyl belinostat/belinostat | 0.0948 (1.53) | 0.112 (1.52) | 0.149 (1.54) | 0.134 (1.38)
  M21/belinostat: number analyzed (Participants) | 14 | 22 | 10 | 15
  M21/belinostat | 0.0522 (1.69) | 0.0642 (1.50) | 0.0768 (1.54) | 0.0759 (1.43)
  M24/belinostat: number analyzed (Participants) | 14 | 22 | 10 | 15
  M24/belinostat | 0.117 (1.36) | 0.0870 (1.61) | 0.0738 (1.46) | 0.0710 (1.84)
  M26/belinostat: number analyzed (Participants) | 14 | 22 | 10 | 15
  M26/belinostat | 0.0752 (1.48) | 0.0666 (1.44) | 0.0824 (1.57) | 0.0806 (1.64)
  M24/M26 | 1.56 (1.46) | 1.32 (1.50) | 0.895 (1.88) | 0.611 (1.66)
  M26/M21 | 1.44 (1.88) | 0.96 (1.62) | 1.07 (1.50) | 1.06 (1.84)
Statistical Analysis 1: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — Belinostat glucuronide/belinostat; p = 0.023, Jonckheere-Terpstra; Kendall's Tau = -0.224
Statistical Analysis 2: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — Methyl belinostat/belinostat; p = 0.011, Jonckheere-Terpstra; Kendall's Tau = 0.295
Statistical Analysis 3: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — M21/belinostat; p = 0.004, Jonckheere-Terpstra; Kendall's Tau = 0.335
Statistical Analysis 4: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — M24/belinostat; p = 0.037, Jonckheere-Terpstra; Kendall's Tau = -0.240
Statistical Analysis 5: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — M26/belinostat; p = 0.275, Jonckheere-Terpstra; Kendall's Tau = 0.127
Statistical Analysis 6: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — M24/M26; p = 0.002, Jonckheere-Terpstra; Kendall's Tau = -0.308
Statistical Analysis 7: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — M26/M21; p = 0.095, Jonckheere-Terpstra; Kendall's Tau = -0.159

11. Primary Outcome: Pharmacokinetics (PK) of Single-dose Belinostat (400 mg/m^2) According to Degree of Liver Dysfunction: Metabolic Ratios of Area Under the Plasma Concentration Time Curve Extrapolated to Infinity (AUC0-inf) for the Belinostat Metabolic Pathway
Description: Metabolic ratios of Area Under the Plasma Concentration Time Curve Extrapolated to Infinity (AUC0-inf), reported as geometric mean (geometric standard deviation), for the belinostat metabolic pathway on Cycle 1 Day-7 as a function of degree of liver dysfunction.
Time Frame: as for outcome 8
Population: The number of patients in a given cohort that received Belinistat on Cycle 1 Day-7 and had blood samples successfully collected at the specified timepoints for PK analysis. One patient with Mild Liver Dysfunction was not evaluable for Belinostat AUC0-inf.
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Normal Function | Mild Dysfunction | Moderate Dysfunction | Severe Dysfunction
Number analyzed (Participants) | 14 | 25 | 10 | 15
ratio
  Belinostat glucuronide/belinostat: number analyzed (Participants) | 14 | 24 | 10 | 15
  Belinostat glucuronide/belinostat | 18.7 (1.63) | 21.8 (1.63) | 18.1 (1.86) | 17.7 (1.91)
  Methyl belinostat/belinostat: number analyzed (Participants) | 14 | 24 | 10 | 15
  Methyl belinostat/belinostat | 0.422 (1.56) | 0.574 (1.53) | 0.892 (1.65) | 0.759 (1.65)
  M21/belinostat: number analyzed (Participants) | 14 | 24 | 10 | 15
  M21/belinostat | 0.901 (3.64) | 0.783 (2.30) | 1.24 (1.85) | 1.13 (2.13)
  M24/belinostat: number analyzed (Participants) | 14 | 24 | 10 | 15
  M24/belinostat | 1.24 (1.55) | 1.01 (1.74) | 0.916 (1.62) | 0.825 (1.96)
  M26/belinostat: number analyzed (Participants) | 14 | 24 | 10 | 15
  M26/belinostat | 0.452 (1.50) | 0.423 (1.49) | 0.666 (1.63) | 0.611 (1.66)
  M24/M26 | 2.74 (1.72) | 2.35 (1.59) | 1.38 (1.91) | 1.35 (2.38)
  M26/M21 | 1.15 (4.14) | 0.531 (2.26) | 0.539 (1.59) | 0.541 (2.63)
Statistical Analysis 1: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — Belinostat glucuronide/belinostat; p = 0.568, Jonckheere-Terpstra; Kendall's Tau = -0.055
Statistical Analysis 2: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — Methyl belinostat/belinostat; p < 0.001, Jonckheere-Terpstra; Kendall's Tau = 0.380
Statistical Analysis 3: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — M21/belinostat; p = 0.001, Jonckheere-Terpstra; Kendall's Tau = 0.315
Statistical Analysis 4: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — M24/belinostat; p = 0.037, Jonckheere-Terpstra; Kendall's Tau = -0.205
Statistical Analysis 5: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — M26/belinostat; p = 0.033, Jonckheere-Terpstra; Kendall's Tau = 0.218
Statistical Analysis 6: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — M24/M26; p = 0.001, Jonckheere-Terpstra; Kendall's Tau = -0.309
Statistical Analysis 7: Comparison: Normal Function vs Mild Dysfunction vs Moderate Dysfunction vs Severe Dysfunction; [analysis description as in outcome 4, analysis 1]; Test type: Other — M26/M21; p = 0.032, Jonckheere-Terpstra; Kendall's Tau = -0.205

12. Secondary Outcome: Best Response
Description: Radiologic response assessments by computed tomography (CT) scans were performed at baseline and every two cycles of treatment based on the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1. Per RECIST v1.1 Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum diameters; Stable Disease (SD), neither sufficient shrinkage to qualify for a PR nor sufficient increase to qualify for Progression of Disease (PD), taking as reference the smallest sum diameters while on study; PD, >=20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study) and an absolute increase of at least 5mm or the appearance of new lesions; Complete Response (CR), Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
Time Frame: at baseline and every two 21-day cycles of treatment, up to 12 cycles
Population: Patients were considered evaluable for response if they received at least one cycle of therapy and had their disease re-evaluated with a restaging scan, or exhibited objective disease progression prior ot the end of Cycle 1 but after receiving all Cycle 1 doses.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Function-Belinostat 1000 mg/m(2) | Mild Dysfunction-Belinostat 750 mg/m(2) | Mild Dysfunction-Belinostat 1000 mg/m(2) | Moderate Dysfunction-Belinostat 500 mg/m(2) | Moderate Dysfunction-Belinostat 750 mg/m(2) | Severe Dysfunction-Belinostat 250 mg/m(2) | Severe Dysfunction-Belinostat 350 mg/m(2)
Number analyzed (Participants) | 14 | 9 | 8 | 4 | 3 | 6 | 3
Participants
  Partial Response | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Stable Disease | 6 | 3 | 1 | 2 | 1 | 0 | 0
  Progressive Disease | 8 | 6 | 7 | 2 | 2 | 6 | 3

13. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0).
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: From Cycle 1 Day -7 up to 12 (21-day) cycles.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Function-Belinostat 1000 mg/m(2) | Mild Dysfunction-Belinostat 750 mg/m(2) | Mild Dysfunction-Belinostat 1000 mg/m(2) | Moderate Dysfunction-Belinostat 500 mg/m(2) | Moderate Dysfunction-Belinostat 750 mg/m(2) | Severe Dysfunction-Belinostat 250 mg/m(2) | Severe Dysfunction-Belinostat 350 mg/m(2)
Number analyzed (Participants) | 14 | 12 | 18 | 5 | 5 | 10 | 8
Participants | 14 | 11 | 14 | 5 | 4 | 9 | 6

ADVERSE EVENTS:
Time Frame: From Cycle 1 Day -7 up to 12 (21-day) cycles.
Arm/Group | Normal Function-Belinostat 1000 mg/m(2) | Mild Dysfunction-Belinostat 750 mg/m(2) | Mild Dysfunction-Belinostat 1000 mg/m(2) | Moderate Dysfunction-Belinostat 500 mg/m(2) | Moderate Dysfunction-Belinostat 750 mg/m(2) | Severe Dysfunction-Belinostat 250 mg/m(2) | Severe Dysfunction-Belinostat 350 mg/m(2)
All-Cause Mortality (participants affected / at risk) | 0/14 | 1/12 | 3/18 | 1/5 | 1/5 | 6/10 | 4/8
Serious Adverse Events (participants affected / at risk) | 5/14 | 6/12 | 7/18 | 4/5 | 3/5 | 7/10 | 4/8
Other Adverse Events (participants affected / at risk) | 14/14 | 11/12 | 14/18 | 5/5 | 4/5 | 9/10 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Function-Belinostat 1000 mg/m(2) (N=14) | Mild Dysfunction-Belinostat 750 mg/m(2) (N=12) | Mild Dysfunction-Belinostat 1000 mg/m(2) (N=18) | Moderate Dysfunction-Belinostat 500 mg/m(2) (N=5) | Moderate Dysfunction-Belinostat 750 mg/m(2) (N=5) | Severe Dysfunction-Belinostat 250 mg/m(2) (N=10) | Severe Dysfunction-Belinostat 350 mg/m(2) (N=8)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 1 (3) | 0 (0) | 3 (3) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (5) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 5 (6) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Function-Belinostat 1000 mg/m(2) (N=14) | Mild Dysfunction-Belinostat 750 mg/m(2) (N=12) | Mild Dysfunction-Belinostat 1000 mg/m(2) (N=18) | Moderate Dysfunction-Belinostat 500 mg/m(2) (N=5) | Moderate Dysfunction-Belinostat 750 mg/m(2) (N=5) | Severe Dysfunction-Belinostat 250 mg/m(2) (N=10) | Severe Dysfunction-Belinostat 350 mg/m(2) (N=8)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (5) | 1 (1) | 1 (1) | 2 (4) | 2 (3) | 0 (0) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 6 (19) | 4 (8) | 3 (6) | 2 (14) | 0 (0) | 3 (4)
Alkaline phosphatase increased (Investigations) | 1 (4) | 3 (7) | 9 (17) | 2 (4) | 2 (3) | 3 (5) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 6 (71) | 4 (7) | 5 (24) | 5 (27) | 2 (3) | 4 (7) | 4 (6)
Anorexia (Metabolism and nutrition disorders) | 3 (43) | 1 (1) | 6 (14) | 3 (7) | 2 (6) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (14) | 1 (8) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 1 (3) | 3 (5) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (6) | 7 (27) | 6 (17) | 2 (4) | 3 (8) | 3 (7) | 4 (7)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (5) | 1 (1) | 0 (0) | 1 (6) | 1 (2) | 1 (2) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 6 (12) | 9 (18) | 5 (17) | 3 (14) | 4 (10) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (2) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (12) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 3 (10) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (14) | 1 (1) | 2 (4) | 1 (2) | 3 (9) | 1 (4) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 2 (6) | 1 (1) | 3 (5) | 2 (3) | 1 (3) | 0 (0) | 2 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (6) | 2 (4) | 2 (4) | 5 (5) | 1 (1) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 3 (13) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dysesthesia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (28) | 3 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (24) | 1 (1) | 3 (5) | 1 (2) | 1 (1) | 0 (0) | 2 (2)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (5) | 4 (8) | 2 (2)
Edema trunk (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 (15) | 2 (2) | 3 (6) | 2 (3) | 0 (0) | 1 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (9) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (23) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophageal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (5) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (12) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 8 (106) | 4 (11) | 7 (14) | 2 (3) | 3 (7) | 2 (3) | 2 (3)
Fever (General disorders) | 2 (3) | 3 (11) | 2 (4) | 3 (16) | 1 (2) | 1 (1) | 1 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 1 (2) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (4) | 3 (12) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (16) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 2 (2) | 2 (2) | 0 | 1 (1) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (8) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (24) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (74) | 1 (16) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (12) | 1 (1) | 2 (11) | 3 (15) | 1 (3) | 0 (0) | 3 (5)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (32) | 4 (7) | 8 (29) | 1 (1) | 2 (3) | 3 (7) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 3 (4) | 1 (3) | 2 (3) | 1 (2) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5) | 6 (8) | 5 (9) | 3 (9) | 1 (2) | 2 (6) | 1 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 2 (9) | 2 (8) | 0 (0) | 2 (7) | 0 | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 4 (26) | 4 (6) | 5 (11) | 3 (12) | 1 (3) | 3 (4) | 3 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 4 (27) | 2 (2) | 3 (6) | 3 (14) | 3 (7) | 2 (2)
Hypotension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 2 (14) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 1 (7) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INR increased (Investigations) | 1 (4) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (9) | 2 (9) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 6 (25) | 3 (4) | 6 (26) | 5 (11) | 0 (0) | 2 (3) | 3 (3)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (50) | 7 (33) | 8 (15) | 5 (13) | 3 (8) | 3 (3) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (55) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (24) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral nerve infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 6 (24) | 2 (4) | 2 (2) | 1 (5) | 2 (2) | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (6) | 2 (2) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 2 (2)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (66) | 0 (0) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (4) | 2 (2) | 3 (4) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (12) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (16) | 6 (24) | 7 (18) | 2 (4) | 2 (4) | 4 (5) | 0
Weight loss (Investigations) | 1 (24) | 0 (0) | 1 (3) | 2 (8) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 2 (15) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT01273155/Prot_SAP_000.pdf
  • Informed Consent Form (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT01273155/ICF_001.pdf